CLINICAL TRIAL: NCT03518619
Title: The Development of a Personalized, Real-time Intervention for Substance-using Emerging Adults Leaving Psychiatric Partial Hospitalization
Brief Title: The Development of a Personalized, Real-time Intervention
Acronym: PFIcope+EMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1803-002; U54GM115677 (NIH)
Record Dates: First submitted 2018-04-25; First posted 2018-05-08 (Actual); Results first posted 2022-11-16 (Actual); Last update posted 2022-11-16 (Actual); Status verified 2022-10

CONDITIONS: Drinking, Alcohol
MeSH Terms: conditions — Alcohol Drinking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PFIcope+EMI (Experimental): This will include: 1) an in-person personalized feedback session to present normative information and feedback on problems associated with drinking to cope, to discuss the individual's use of alcohol to cope, and to generate relapse prevention coping skills messages to be used in the EMI text intervention; 2) EMA to monitor affect and intention to drink after discharge; 3) tailored text messages (EMI) based on EMA responses (i.e., individualized coping skills messages when individuals report negative affect and intention to drink); and 4) additional EMA to monitor coping skills usage, alcohol use, and drinking to cope.
  Interventions: Behavioral: PFIcope+EMI

INTERVENTIONS:
Behavioral: PFIcope+EMI — The intervention will be comprised of (1) an initial orientation session where the intervention is introduced, receipt of personalized normative information, motives feedback, and the development of an individual's personalized relapse prevention coping skills messages to be utilized through the course of the intervention; (2) EMA for monitoring of affect, drinking intention, alcohol use, and coping skills use; (3) EMI-tailored text messages sent based on EMA responses: individualized, self-chosen relapse prevention coping skills messages when participants report negative affect and intent to drink.

SUMMARY:
The investigators propose to enhance our existing coping motive-specific normative feedback intervention (PFIcope intervention) by capitalizing on EMA/EMI technology to pair real-time affective monitoring with tailored real-time relapse prevention texts for individuals with anxiety and depression who drink to cope. The goals of the PFIcope+EMI study are to help individuals to identify motives for drinking and to utilize alternate coping strategies for negative affect in place of alcohol.

DETAILED DESCRIPTION:
Emerging adulthood (ages 18-25) represents and common and problematic time for alcohol use and mental health issues, particularly anxiety and depression. Anxiety and depression increase the likelihood of developing risky patterns of alcohol use. Indeed, individuals who drink alcohol to cope with negative affect, such as anxiety and depression, report more alcohol use and more severe use-related consequences. As such, it is important to address alcohol use, particularly among a psychiatric population of emerging adults. Despite their co-occurrence, treatment as usual for anxiety and depression typically does not address alcohol use, and alcohol interventions for emerging adults largely ignore anxiety and depression. Emerging research suggests interventions that specifically focus on drinking to cope with negative affect are promising in reducing problematic outcomes. For example, the investigators previously developed a brief, personalized feedback intervention that specifically targeted use of alcohol to cope with negative affect among a normative sample of emerging adults (Personalized Feedback Intervention for Coping - PFIcope), which resulted in decreased drinking to cope. In order to adapt PFIcope for a psychiatric population and augment treatment effects, the investigators propose adding ecological momentary assessment (EMA) and intervention (EMI) in order to identify when emerging adults are at most risk for problematic alcohol use and intervene when needed. EMA can assess symptoms in real time and identify high-risk situations for problematic use (i.e., when experiencing negative affect and reports intention to use), which can trigger an in-the-moment EMI during that high-risk situation (i.e., individually-chosen relapse prevention coping skills messages).

The investigators propose to develop a 6-week PFIcope+EMI intervention for 20 emerging adults in a psychiatric partial hospitalization program who report drinking alcohol to cope with negative affect. This will include: 1) an in-person personalized feedback session to present normative information and feedback on problems associated with drinking to cope, to discuss the individual's use of alcohol to cope, and to generate relapse prevention coping skills messages to be used in the EMI text intervention; 2) EMA to monitor affect and intention to drink after discharge; 3) tailored text messages (EMI) based on EMA responses (i.e., individualized coping skills messages when individuals report negative affect and intention to drink); and 4) additional EMA to monitor coping skills usage, alcohol use, and drinking to cope. The PFIcope+EMI intervention, including its associated real-time assessment and messaging systems, is low-cost, easy to program, and can deliver an intervention when individuals are at most risk for engaging in problematic alcohol use.

ELIGIBILITY:
Inclusion Criteria:

(a) between 18 and 25 years of age, (b) reported alcohol use at least 3x weekly over past month, (c) self-reported use of coping motive (mean of 2+ on coping subscale of MDMQ-R), (d) current anxiety and/or depression symptomatology (as assessed CES-D score of 16+ and GAD-7 scores 10+), (e) has access to a smartphone capable of receiving EMA and text, and access to email.

Exclusion Criteria:

(a) current DSM-5 diagnosis of moderate/severe other substance use disorder (i.e., other than alcohol), (b) a history of psychotic disorder or current psychotic symptoms, (c) current suicidal/homicidal ideation.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2018-09-24 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from a Young Adult Partial Hospitalization program at a private psychiatric institution. Recruitment occurred between September 2018 and February 2019.
Period: Overall Study
Arm/Group | PFIcope+EMI
Started | 20
Completed | 15
Not Completed | 5

BASELINE CHARACTERISTICS:
Population: After the baseline, 5 participants decided not to participate in the intervention.
Arm/Group | PFIcope+EMI
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.74 (2.23)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 17
  More than one race | 1
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 20
Percent Days Drinking [Mean (Standard Deviation); unit: Percentage of days] — Percent of days over the last 90 days where a participant endorsed drinking alcohol. This data was collected using the Timeline Followback Interview.
  Percentage of days | 35 (25)
Drinks per Drinking Day (DDD) [Mean (Standard Deviation); unit: alcoholic drinks] — Over the last 90 days, on days when the participant drank alcohol, the mean number of drinks that were consumed. This data was obtained from the Timeline Followback Interview.
  alcoholic drinks | 3.56 (1.67)
Percent Days Binge Drinking [Mean (Standard Deviation); unit: Percentage of days] — The percent of days in the last 90 days when a participant engaged in binge drinking. Binge drinking is defined as 4 or more drinks in a single episode for women and 5 or more drinks in a single episode for a male. Data was collected using the Timeline Followback Interview.
  Percentage of days | 21.70 (8.25)
Social Drinking Motives [Mean (Standard Deviation); unit: units on a scale] — Alcohol use motives were measured using the Modified Drinking Motives Questionnaire-Revised. Social drinking motives are a subscale of this measure. The subscale items range from 1=Almost Never/Never to 5=Almost Always/Always. Subscale scores reflect the mean of items. Higher values reflect drinking for social motives.
  units on a scale | 3.3 (0.43)
Coping with Anxiety Drinking Motives [Mean (Standard Deviation); unit: units on a scale] — Alcohol use motives were measured using the Modified Drinking Motives Questionnaire-Revised. Coping with anxiety drinking motives are a subscale of this measure. The subscale items range from 1=Almost Never/Never to 5=Almost Always/Always. Subscale scores reflect the mean of items. Higher values reflect drinking for coping with anxiety.
  units on a scale | 3.42 (1.14)
Coping with Depression Drinking Motives [Mean (Standard Deviation); unit: units on a scale] — Alcohol use motives were measured using the Modified Drinking Motives Questionnaire-Revised. Coping with depression drinking motives are a subscale of this measure. The subscale items range from 1=Almost Never/Never to 5=Almost Always/Always. Subscale scores reflect the mean of items. Higher values reflect drinking for coping with depression motives.
  units on a scale | 2.85 (1.49)
Enhancement Drinking Motives [Mean (Standard Deviation); unit: units on a scale] — Alcohol use motives were measured using the Modified Drinking Motives Questionnaire-Revised. Enhancement drinking motives are a subscale of this measure. The subscale items range from 1=Almost Never/Never to 5=Almost Always/Always. Subscale scores reflect the mean of items. Higher values reflect drinking for enhancement motives.
  units on a scale | 3.37 (0.93)
Conformity Drinking Motives [Mean (Standard Deviation); unit: units on a scale] — Alcohol use motives were measured using the Modified Drinking Motives Questionnaire-Revised. Conformity drinking motives are a subscale of this measure. The subscale items range from 1=Almost Never/Never to 5=Almost Always/Always. Subscale scores reflect the mean of items. Higher values reflect drinking for conformity motives.
  units on a scale | 1.6 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: Drinking Motives Questionnaire-Revised (DMQ-R) Coping Motive
Description: Drinking to cope with negative affect, 5 items on scale of 1-5 with higher values meaning more use
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PFIcope+EMI
Number analyzed (Participants) | 15
score on a scale | 2.15 (.82)
Statistical Analysis 1: Comparison: PFIcope+EMI; Test type: Other — This is a single group design. Paired-samples t-tests were conducted; p < .05, t-test, 2 sided — This is a calculated p-value

2. Primary Outcome: Percentage of Days of Alcohol Use in the Last Month
Description: Alcohol use, yes/no for each day of past 30
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: percentage of drinking days
Arm/Group | PFIcope+EMI
Number analyzed (Participants) | 15
percentage of drinking days | 19 (22)
Statistical Analysis 1: Comparison: PFIcope+EMI; Test type: Other — This is a single group design. Paired-samples t-tests were conducted; p < .01, t-test, 2 sided — This is a calculated p-value

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: It does not differ from clinicaltrials.gov
Arm/Group | PFIcope+EMI
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 2/20
Other Adverse Events (participants affected / at risk) | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PFIcope+EMI (N=20)
Psychiatric Inpatient Hospitalization (Psychiatric disorders) | 2 (2) — The participant was psychiatrically hospitalized during the 6-week intervention.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03518619/Prot_SAP_000.pdf
  • Informed Consent Form (2021-01-15): https://cdn.clinicaltrials.gov/large-docs/19/NCT03518619/ICF_001.pdf